CLINICAL TRIAL: NCT05399641
Title: Oral Ibrexafungerp for the Treatment of Complicated Vulvovaginal Candidiasis (VVC) in Subjects Who Have Failed Fluconazole Therapy
Brief Title: Ibrexafungerp for the Treatment of Complicated Vulvovaginal Candidiasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCY-078-307b
Record Dates: First submitted 2022-05-23; First posted 2022-06-01 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Vulvovaginal Candidiasis
Keywords: vulvovaginal candidiasis; candida; VVC; rVVC; Ibrexafungerp; yeast vaginitis
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Torulopsis | interventions — ibrexafungerp

STUDY DESIGN:
Intervention Model Description: Open-label, 3 group, stratified
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Subjects without underlying medical conditions and have isolates other than C glabrata, C krusei, C auris.
  Single day dosing, 300mg Ibrexafungerp BID for a total of 600mg a day.
  Interventions: Drug: Ibrexafungerp
- Group B (3 Day dosing) (Experimental): Subjects with underlying medical conditions: DM, immunocompromised conditions (e.g. HIV), debilitation, immunosuppressive therapy (e.g. corticosteroids), recurrent VVC (≥3 episodes/year) and/or known to have C glabrata, C krusei or C auris isolates.
  Three day dosing, 300 mg Ibrexafungerp BID for a total of 600mg a day.
  Interventions: Drug: Ibrexafungerp
- Group B (7 Day dosing) (Experimental): Subjects with underlying medical conditions: DM, immunocompromised conditions (e.g. HIV), debilitation, immunosuppressive therapy (e.g. corticosteroids), recurrent VVC (≥3 episodes/year) and/or known to have C glabrata, C krusei or C auris isolates.
  Seven day dosing, 300mg Ibrexafungerp BID for a total of 600mg a day
  Interventions: Drug: Ibrexafungerp

INTERVENTIONS:
Drug: Ibrexafungerp — Each day dosing will consist of two 150mg tablets taken BID.

SUMMARY:
This study will treat subjects with complicated VVC who have failed prior fluconazole therapy with Ibrexafungerp for 1, 3 or 7 days of treatment.

DETAILED DESCRIPTION:
This study will treat subjects with complicated VVC who have failed prior fluconazole therapy with Ibrexafungerp for 1, 3 or 7 days of treatment.

Approximately 150 eligible subjects will be enrolled. Subjects will be randomized to receive oral ibrexafungerp 300 mg administered twice a day (BID) for either one, three, or seven consecutive days, stratified by group based on Candida species and presence or absence of underlying medical conditions.

The primary endpoint for this study is the percentage of subjects with a clinical cure at the Test of Cure Visit. Test of Cure is defined as a score of zero on the Vulvovaginal Signs and Symptoms Scale and not requiring additional antifungal treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a post menarchal female ≥18 years of age at the time of signing the ICF.
2. Subject has a diagnosis of symptomatic VVC that meets the following criteria at the

   Screening visit:
   1. Minimum composite vulvovaginal signs and symptoms score of ≥4 with at least 2 signs or symptoms having a score of 2 (moderate) or greater on the VSS scale at baseline.
   2. Positive microscopic examination with 10% KOH in a vaginal sample collected at Screening revealing yeast forms (hyphae/pseudohyphae) or budding yeasts
   3. Normal vaginal pH (≤ 4.5).
   4. Has no other vaginal co-infections based on wet mount microscopic examination (and/or DNA probe).
3. Subject should also have:

   1. A VVC with persistent symptoms despite fluconazole therapy (last dose of fluconazole must have been administered at least 7 days prior, but no longer than 28 days prior to screening. OR
   2. A recurrent vulvovaginal candidiasis (RVVC) episode with breakthrough symptoms while receiving maintenance antifungal therapy. OR
   3. A VVC episode caused by a non-albicans candida species known to have either intrinsic resistance to fluconazole e.g. C.krusei or suspected resistance to fluconazole, e.g. C.glabrata, C. auris but likely without MIC data in hand. OR
   4. A VVC episode caused by Candida species with documented resistance to fluconazole based on MIC determination. OR
   5. A known history of azole allergy or intolerance.
4. Subject is able to take oral tablets.
5. Subject is not pregnant or lactating and plans not to become pregnant. Women of childbearing potential < 1 year post-menopausal must agree to and comply with using one barrier method (male condom, female condom, and diaphragm) plus one other highly effective method of birth control, or sexual abstinence, from the time of consent through 10 days after the completion of study therapy. Subjects must refrain from using any topical vaginal contraceptives as these may have an impact on the signs and symptoms of VVC. Note: Women of childbearing potential must have a negative urine pregnancy test prior to enrollment (performed by the site's local laboratory).
6. Subject is able to understand and sign a written ICF, which must be obtained prior to treatment and any study-related procedures.
7. Subject is able to understand and sign a consent or authorization form, which shall permit the use, disclosure and transfer of the subject's personal health information (e.g., in the US Health Information Portability and Accountability Act Authorization form).
8. Subject is able to understand and follow all study-related procedures including study drug administration.

Exclusion Criteria:

1. Subject has any vaginal condition other than VVC that may interfere with the diagnosis or evaluation of response to therapy, such as concurrent causes of vulvovaginitis and/or cervicitis including bacterial vaginosis, Trichomonas, Herpes virus, Neisseria gonorrhoeae, Chlamydia, symptomatic human papillomavirus infection, or other mixed infections.
2. Subject received systemic and/or topical vaginal antifungal treatment, including prescription or over-the-counter products, within 7 days prior to the Screening visit.

   Note: The screening visit may be rescheduled if required.
3. Subject is receiving or anticipates requiring treatment with the prohibited medications within the specified timeframes per Appendix I.
4. Subject has active menstruation at the Screening visit. Note: The Screening visit may be rescheduled if required.
5. Subject has a history of or an active cervical/vaginal cancer.
6. Subject has a known hypersensitivity to any of the components of the formulation.
7. Subject has participated in any other investigational study within at least 30 days (or 5.5 half- lives of the investigational product) before signing the ICF.
8. Subject has received prior treatment with ibrexafungerp.
9. Subject has any other condition or laboratory abnormality (such as severe hepatic impairment) that, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study or may interfere with the assessments included in the study.
10. Subject is unlikely to comply with protocol requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Tierney, Study Director — Scynexis, Inc.
Locations (25):
- United States (25):
  - Precision Trials, AZ, Phoenix, Arizona
  - Women's Healthcare Research, San Diego, California
  - Wake Research (MCCR), San Diego, California
  - New Age Medical Research, Miami, Florida
  - Wake (Mount Vernon Clinical Research), Atlanta, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Leavitt Women's Healthcare, Idaho Falls, Idaho
  - Women Under Study, New Orleans, Louisiana
  - Massachusetts's General, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Consultants in Women's Healthcare, St Louis, Missouri
  - Wake Research (CRCN), Las Vegas, Nevada
  - Capital Health Lawrence OBGYN, Lawrenceville, New Jersey
  - Center for Colposcopy, Lake Success, New York
  - Wake Research (Carolina Institute for Clinical Research), Fayetteville, North Carolina
  - UWCR - Raleigh, Raleigh, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Jefferson University, Philadelphia, Pennsylvania
  - Medical Research Center, Memphis, Tennessee
  - Discovery Clinical Trials, Dallas, Texas
  - TMC Life Research, Inc, Houston, Texas
  - Discovery Clinical Trials, McAllen, Texas
  - Seattle Clinical Research Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Single day dosing, 300mg Ibrexafungerp BID for a total of 600mg a day.
  Ibrexafungerp: Each day dosing will consist of two 150mg tablets taken BID.
- Group B (3 Day Dosing): Three day dosing, 300 mg Ibrexafungerp BID for a total of 600mg a day.
  Ibrexafungerp: Each day dosing will consist of two 150mg tablets taken BID.
- Group B (7 Day Dosing): Seven day dosing, 300mg Ibrexafungerp BID for a total of 600mg a day
  Ibrexafungerp: Each day dosing will consist of two 150mg tablets taken BID.
Period: Overall Study
Arm/Group | Group A | Group B (3 Day Dosing) | Group B (7 Day Dosing)
Started | 27 | 62 | 61
Completed | 18 | 40 | 42
Not Completed | 9 | 22 | 19
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Physician Decision | 1 | 3 | 3
Not completed — Withdrawal by Subject | 4 | 11 | 7
Not completed — Reason not defined | 3 | 5 | 6

BASELINE CHARACTERISTICS:
Population: Intent- to Treat Set (ITT) - all ibrexafungerp-treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B (3 Day Dosing) | Group B (7 Day Dosing) | Total
Number analyzed (Participants) | 27 | 62 | 61 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (14.80) | 39.6 (13.50) | 39.3 (11.43) | 39.6 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 62 | 61 | 150
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 14 | 18 | 38
  Not Hispanic or Latino | 21 | 48 | 43 | 112
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 3 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 15 | 14 | 40
  White | 13 | 42 | 45 | 100
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure
Description: Percentage of participants with complete resolution of signs and symptoms (total VSS score of 0) with no additional antifungal therapy required. The vulvovaginal signs and symptom (VSS) scale ranges from 0 to 18, with higher scores being worse.
Time Frame: 14 days post-Baseline - Test-Of-Cure (TOC)
Population: Modified Intent-to-Treat (mITT): all treated participants who have a positive culture for candida species at screening
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B (3 Day Dosing) | Group B (7 Day Dosing)
Number analyzed (Participants) | 13 | 42 | 46
Participants | 7 | 10 | 23

2. Secondary Outcome: Clinical Improvement
Description: Percentage of participants with a Total Composite Score of ≤1 on the VSS Scale and a Total Composite Score of ≤2 on the VSS scale. The vulvovaginal signs and symptom (VSS) scale ranges from 0 to 18, with higher scores being worse.
Time Frame: 14 days post-Baseline Test-Of- Cure (TOC), 14 days post-End of Treatment (EOT), 30 days post-Baseline, 30 days post-End of Treatment and 60 days post-End of Treatment
Population: Modified Intent-to-Treat (mITT): all treated participants who have a positive culture for candida species at screening
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B (3 Day Dosing) | Group B (7 Day Dosing)
Number analyzed (Participants) | 13 | 42 | 46
Participants
  VSS Score ≤1, (TOC) | 10 | 20 | 29
  VSS Score ≤2, (TOC) | 11 | 23 | 33
  VSS Score ≤1, (14 days post-EOT): number analyzed (Participants) | 3 | 15 | 34
  VSS Score ≤1, (14 days post-EOT) | 3 | 8 | 22
  VSS Score ≤1, (30 days post-Baseline): number analyzed (Participants) | 12 | 31 | 33
  VSS Score ≤1, (30 days post-Baseline) | 10 | 18 | 24
  VSS Score ≤1, (30 days post-EOT: number analyzed (Participants) | 3 | 11 | 26
  VSS Score ≤1, (30 days post-EOT | 3 | 8 | 20
  VSS Score ≤1, (60 days post-EOT): number analyzed (Participants) | 9 | 21 | 28
  VSS Score ≤1, (60 days post-EOT) | 8 | 18 | 21
  VSS Score ≤2, (14 days post-EOT): number analyzed (Participants) | 3 | 15 | 34
  VSS Score ≤2, (14 days post-EOT) | 3 | 10 | 26
  VSS Score ≤2, (30 days post-Baseline): number analyzed (Participants) | 12 | 31 | 33
  VSS Score ≤2, (30 days post-Baseline) | 10 | 20 | 26
  VSS Score ≤2, (30 days post-EOT): number analyzed (Participants) | 3 | 11 | 26
  VSS Score ≤2, (30 days post-EOT) | 3 | 8 | 20
  VSS Score ≤2, (60 days post-EOT): number analyzed (Participants) | 9 | 21 | 28
  VSS Score ≤2, (60 days post-EOT) | 8 | 18 | 24

3. Secondary Outcome: Clinical Success
Description: Percentage of participants with at least 50% reduction from baseline in the total composite VSS score and no additional antifungal therapy required. The vulvovaginal signs and symptom (VSS) scale ranges from 0 to 18, with higher scores being worse.
Time Frame: as for outcome 2
Population: Modified Intent-to-Treat (mITT): all treated participants who have a positive culture for candida species at screening
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B (3 Day Dosing) | Group B (7 Day Dosing)
Number analyzed (Participants) | 13 | 42 | 46
Participants
  TOC | 11 | 31 | 39
  14 days post-EOT: number analyzed (Participants) | 3 | 15 | 34
  14 days post-EOT | 3 | 12 | 28
  30 days post-Baseline: number analyzed (Participants) | 12 | 31 | 33
  30 days post-Baseline | 10 | 23 | 27
  30 days post-EOT: number analyzed (Participants) | 3 | 11 | 26
  30 days post-EOT | 3 | 9 | 22
  60 days post-EOT: number analyzed (Participants) | 9 | 21 | 28
  60 days post-EOT | 8 | 18 | 25

4. Secondary Outcome: Mycological Response
Description: Percentage of participants with negative culture growth for candida or participant was asymptomatic and a culture was not done
Time Frame: as for outcome 2
Population: Modified Intent-to-Treat (mITT): all treated participants who have a positive culture for candida species at Screening
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B (3 Day Dosing) | Group B (7 Day Dosing)
Number analyzed (Participants) | 13 | 42 | 46
Participants
  TOC | 9 | 23 | 31
  14 days post-EOT: number analyzed (Participants) | 3 | 15 | 34
  14 days post-EOT | 3 | 8 | 21
  30 days post-Baseline: number analyzed (Participants) | 12 | 31 | 32
  30 days post-Baseline | 7 | 18 | 25
  30 days post-EOT: number analyzed (Participants) | 3 | 11 | 26
  30 days post-EOT | 3 | 9 | 20
  60 days post-EOT: number analyzed (Participants) | 9 | 21 | 28
  60 days post-EOT | 9 | 19 | 24

5. Secondary Outcome: Clinical Cure and Mycological Response
Description: The number (percentage) of participants with Clinical Cure and Mycological Response at TOC and FU Visits
Time Frame: as for outcome 2
Population: Modified Intent-to-Treat (mITT) - all treated participants who have a positive culture for candida species at Screening
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B (3 Day Dosing) | Group B (7 Day Dosing)
Number analyzed (Participants) | 13 | 42 | 46
Participants
  TOC | 5 | 7 | 16
  14 days post-EOT: number analyzed (Participants) | 3 | 15 | 34
  14 days post-EOT | 3 | 5 | 13
  30 days post-Baseline: number analyzed (Participants) | 12 | 31 | 32
  30 days post-Baseline | 7 | 15 | 20
  30 days post-EOT: number analyzed (Participants) | 3 | 11 | 26
  30 days post-EOT | 3 | 8 | 17
  60 days post-EOT: number analyzed (Participants) | 9 | 21 | 28
  60 days post-EOT | 8 | 17 | 20

6. Secondary Outcome: Clinical Cure at Follow-up
Description: The number (percentage) of participants with a total composite score of 0 on the VSS scale and no additional antifungal therapy required. The vulvovaginal signs and symptom (VSS) scale ranges from 0 to 18, with higher scores being worse.
Time Frame: 14 days post EOT, 30 days post-Baseline, 30 days post-EOT and 60 days post-EOT
Population: Modified Intent-to-Treat (mITT): all treated participants who have a positive culture for candida species at Screening
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B (3 Day Dosing) | Group B (7 Day Dosing)
Number analyzed (Participants) | 13 | 42 | 46
Participants
  14 days post-EOT: number analyzed (Participants) | 3 | 15 | 34
  14 days post-EOT | 3 | 6 | 17
  30 days post-Baseline: number analyzed (Participants) | 12 | 31 | 33
  30 days post-Baseline | 7 | 16 | 21
  30 days post-EOT: number analyzed (Participants) | 3 | 11 | 26
  30 days post-EOT | 3 | 8 | 17
  60 days post-EOT: number analyzed (Participants) | 9 | 21 | 28
  60 days post-EOT | 8 | 17 | 20

7. Secondary Outcome: Change in Total Composite Vulvovaginal Signs and Symptom Score From Baseline
Description: The mean change in total composite vulvovaginal signs and symptom (VSS) score from Baseline to TOC and Follow-up Visits. The VSS score ranges from 0 (no signs and symptoms) to a maximum of 18, with higher scores being worse.
Time Frame: From Baseline to 14 days post-Baseline (TOC), 14 days post-End of Treatment (EOT), 30 days post-Baseline, 30 days post-EOT and 60 days post-EOT
Population: Modified Intent-to-Treat (mITT): all treated participants who have a positive culture for candida species at Screening
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Group A | Group B (3 Day Dosing) | Group B (7 Day Dosing)
Number analyzed (Participants) | 13 | 42 | 46
Score on a scale
  TOC | -7.2 [-15 to 0] | -6.3 [-13 to 4] | -8.1 [-16 to 2]
  14 days post-EOT: number analyzed (Participants) | 3 | 15 | 34
  14 days post-EOT | -10.0 [-11 to -8] | -6.7 [-14 to 2] | -7.8 [-16 to 4]
  30 days post-Baseline: number analyzed (Participants) | 12 | 31 | 33
  30 days post-Baseline | -7.0 [-17 to 9] | -7.1 [-13 to 3] | -8.3 [-17 to 5]
  30 days post-EOT: number analyzed (Participants) | 3 | 11 | 26
  30 days post-EOT | -10.7 [-11 to -10] | -7.6 [-13 to 0] | -8.0 [-16 to 9]
  60 days post-EOT: number analyzed (Participants) | 9 | 21 | 28
  60 days post-EOT | -8.3 [-17 to -3] | -8.2 [-16 to 2] | -8.5 [-16 to 2]

8. Secondary Outcome: Clinical Improvement - 2
Description: Percentage of subjects with a Total Composite Score of 2 on the VSS Scale or a composite score of 1 on the VSS scale. The vulvovaginal signs and symptom (VSS) scale ranges from 0 to 18, with higher scores being worse.
Time Frame: 14 days post-Baseline Test-Of- Cure (TOC), 14 days post-End of Treatment, 30 days post-Baseline, 30 days post-End of Treatment and 60 days post- End of Treatment
Population: Modified Intent-to-Treat (mITT): all treated participants who have a positive culture for candida species at Screening
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B (3 Day Dosing) | Group B (7 Day Dosing)
Number analyzed (Participants) | 13 | 42 | 46
Participants
  VSS Score of 1 at TOC | 3 | 10 | 6
  VSS Score of 1 at 14 days post-EOT: number analyzed (Participants) | 3 | 15 | 34
  VSS Score of 1 at 14 days post-EOT | 0 | 2 | 5
  VSS Score of 1 at 30 days post-Baseline: number analyzed (Participants) | 12 | 31 | 33
  VSS Score of 1 at 30 days post-Baseline | 3 | 2 | 3
  VSS Score of 1 at 30 days post-EOT: number analyzed (Participants) | 3 | 11 | 26
  VSS Score of 1 at 30 days post-EOT | 0 | 0 | 3
  VSS Score of 1 at 60 days post-EOT: number analyzed (Participants) | 9 | 21 | 28
  VSS Score of 1 at 60 days post-EOT | 0 | 1 | 1
  VSS Score of 2 at TOC | 1 | 3 | 4
  VSS Score of 2 at 14 days post-EOT: number analyzed (Participants) | 3 | 15 | 34
  VSS Score of 2 at 14 days post-EOT | 0 | 2 | 4
  VSS Score of 2 at 30 days post-Baseline: number analyzed (Participants) | 12 | 31 | 33
  VSS Score of 2 at 30 days post-Baseline | 0 | 2 | 2
  VSS Score of 2 at 30 days post-EOT: number analyzed (Participants) | 3 | 11 | 26
  VSS Score of 2 at 30 days post-EOT | 0 | 0 | 0
  VSS Score of 2 at 60 days post-EOT: number analyzed (Participants) | 9 | 21 | 28
  VSS Score of 2 at 60 days post-EOT | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: From participant Screening through to 60 post-End of Therapy Visit (approximately 69 days after Screening)
Arm/Group | Group A | Group B (3 Day Dosing) | Group B (7 Day Dosing)
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/62 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/62 | 0/61
Other Adverse Events (participants affected / at risk) | 12/27 | 35/62 | 39/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=27) | Group B (3 Day Dosing) (N=62) | Group B (7 Day Dosing) (N=61)
Diarrhoea (Gastrointestinal disorders) | 6 | 18 | 20
Nausea (Gastrointestinal disorders) | 3 | 16 | 7
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 3 | 4
Constipation (Gastrointestinal disorders) | 0 | 1 | 5
Bacterial vaginosis (Gastrointestinal disorders) | 3 | 1 | 5
Headache (Gastrointestinal disorders) | 1 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT05399641/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT05399641/SAP_001.pdf